CLINICAL TRIAL: NCT07059442
Title: Screening for Anal Cancer and Precancer in Women With HIV (SANCA)
Acronym: SANCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Stockholm South General Hospital (Other); Sahlgrenska University Hospital (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Christina Carlander, PI, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-06554
Record Dates: First submitted 2025-06-13; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Anal Canal Cancer
Keywords: HIV; Human papilloma virus; DNA methylation
MeSH Terms: conditions — Anal Canal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anal HPV testing (Other): All included women will leave an anal HPV-self test
  Interventions: Diagnostic Test: anal HPV screening

INTERVENTIONS:
Diagnostic Test: anal HPV screening — From all included women samples will be collected at the out-patient HIV departments including self-sampled vaginal swab for hrHPV testing and self-sampled anal swab for hrHPV. A blood sample will be taken for the analysis of circulating HPV DNA.

SUMMARY:
The main aim of the SANCA study is to evaluate the feasibility, cost-effectiveness, and acceptability of implementing international anal cancer screening guidelines for women living with HIV in Sweden, integrating health economic and patient-centered approaches.

Secondly the investigators wish to investigate the predictive potential of DNA methylation markers for the clinical progression of precancerous anal lesions in women with HIV, combining prospective molecular biology analysis with clinical data from registries.

DETAILED DESCRIPTION:
Aims and purposes:

(I) Evaluate the feasibility, cost-effectiveness, and acceptability of implementing international anal cancer screening guidelines for women living with HIV in Sweden, integrating health economic and patient-centered approaches.

(II) Assess the combination of Human Papilloma Virus (HPV) type and HPV ct values as a tool for stratifying clinical management (II) Investigate the predictive potential of DNA methylation markers for the clinical progression of precancerous anal lesions in women with HIV (III) Assess circulating HPV DNA in plasma as a highly specific pre-diagnostic biomarker for anal cancer

SUB PROJECT A Study design: Prospective register-based cohort study Study population: All women with HIV from the age of 45 attending routine appointments at the out-patient HIV departments at Karolinska University Hospital in Stockholm (n=707), the South Hospital in Stockholm (n=163), and Sahlgrenska University Hospital in Gothenburg (n=188), Sweden. Patients that fill the inclusion criteria will be identified from the National HIV registry InfCareHIV.

Overall aim: To assess if anal cancer screening, as proposed by the International Anal Neoplasia Society, is feasible (i.e. practical, acceptable, cost-effective) in women 45+ living with HIV Specific research questions

* Which HPV genotypes are seen in anal compared to vaginal self-tests?
* What is the correlation between self-sampled vaginal HPV and self-sampled anal HPV?
* Can the combination of HPV type and cycle threshold HPV levels be used to triage the follow-up of women with HIV that have positive anal hrHPV tests?
* Can circulating HPV DNA (plasma) be used to predict which individuals will develop anal cancer and precancer?
* What is the correlation between hrHPV, anal cytology results and biopsy-results?
* What risk factors are identified for HSIL
* What is the burden of HSIL in women given the level of immunosuppression (severe immunosuppression defined as CD4 count <200)?
* Which HPV genotypes are seen post treatment of anal lesions & post HPV vaccination
* Is anal cancer screening acceptable by women included in the study?
* Is anal cancer screening cost-effective in women 45+ living with HIV? Inclusion: All individuals with a cervix 45+ years living with HIV attending routine appointments at the out-patient HIV departments at Karolinska University Hospital in Stockholm, the South Hospital in Stockholm, and Sahlgrenska University Hospital in Gothenburg, will be asked to give written consent to be included in the study . Information about the study will be given orally and written (Easy Swedish and English). Women that cannot understand Swedish or English will be informed about the study with the help of an interpreter. Written information will be accessible in Swedish, English, Russian, Arabic, Tigrinja, Swahili, Thai, Amharic, and Somali. This is important given that 70% of women with HIV in Sweden were born outside Sweden. Exclusion: Women who have had a rectal amputation will be excluded.

Reject log: data of women who reject inclusion Data collection: Samples will be collected at the out-patient HIV department including self-sampled vaginal swab for hrHPV testing and self-sampled anal swab for hrHPV. A blood sample will be taken for the analysis of circulating HPV DNA. Participants with positive anal hrHPV test will be referred to flexible endoscopy at Ersta diakoni (for women in Stockholm region) or HRA at the Gynecology department at Sahlgrenska University Hospital (for women in Gothenburg region) for anal cytology, anal biopsy and samples for DNA methylation markers. Treatment will be given if needed according to clinical practice. Participants with positive vaginal hrHPV will be referred to gynecologist according to clinical practice. A Case Report Form will be filled in by the research nurses and registered in Red-Cap. Demographic and clinical data will be collected from InfCareHIV and from medical records (history of cervical-, vaginal-, or vulval-dysplasia and comorbidities).

Questionnaire: The participants will answer a questionnaire (level of education, employment, sexual history, smoking) and questions on the acceptability of screening. The questionnaire will be answered by the patient online (using personal mobile phone or research I-pad), recorded with a unique study-id and automatically imported to Red-Cap. The health personnel will not have access to the answers of the questionnaires, but the health personnel will support the participants with any concerns before and after study inclusion.

HPV vaccination: All women that are treated for anal and cervical precancerous lesions within the frame of this study will be offered HPV vaccinations.

Bio bank: The swab samples and biopsies will be stored according to clinical routine in the Stockholm region biobank. The samples are managed according to the Swedish Biobanks in Medical Care Act (2023:38).

Laboratory analysis of circulating HPV DNA: Circulating HPVDNA in plasma will be measured using a digital PCR assay. Circulating HPVDNA will be isolated from 995 μl of plasma using the MP96 DNA and Viral NA Large Volume Kit with the cfNA ss 2000 protocol on the Roche MagNA Pure 96 system. Isolated circulating HPVDNA (and control human beta-globin gene) will be analyzed by a dPCR protocol.

Data analysis and statistics. Statistical analysis: Descriptive analysis will used to describe the study population and chi-square tests for categorical variables and t-tests for continuous variables will be used to compare the prevalence of hrHPV, LSIL and HSIL between subgroups (e.g. based on lowest CD4 count). Multivariable logistic regression will be used to identify factors associated with the presence of HSIL, adjusted for possible confounders such as age and smoking. The investigators will test for trends in sensitivity and specificity of circulating HPVDNA across time windows prior to HSIL/anal cancer diagnosis using logistic regression models. Power calculation: A sample size of 150-300 women will provide the investigators with 80% statistical power (assuming α=0.05) given an expected prevalence of anal hrHPV between 30-60%.Cost-effectiveness analysis will be performed assessing the medical costs for screening in comparison with the medical costs following an anal cancer diagnosis. The medical costs will include direct screening costs, follow-up and treatment costs and indirect costs such as loss of productivity. The time horizon for the analysis will be a lifetime. The primary effectiveness measure will be the number of cases of anal cancer prevented due to screening and early treatment of HSIL. Secondary outcomes will include the number of HSIL cases detected and treated, and quality-adjusted life years gained from preventing cancer progression. Using a decision tree or Markov model the investigators will simulate the natural history of anal cancer in women with HIV. The model will include different health states (e.g. no HSIL, HSIL, early-stage anal cancer, late-stage anal cancer) and transitions between these states based on screening and treatment. The Incremental Cost-effectiveness Ratio (ICER) will be calculated and expressed as cost per quality-adjusted life years or by cancer case prevented. Sensitivity analyses will be performed to test the robustness of the model. A cost-effectiveness threshold will be determined and assessment of whether the screening strategy falls below this threshold, indicating that it is cost-effective.

SUB PROJECT B Study design: Prospective register-based cohort study Study population: All women with HIV included in sub project A that were referred to HRA/flexible endoscopy.

Research questions:

1. Can self-sampled host DNA methylation markers be used for triaging the follow-up of women with HIV that have positive anal hrHPV tests?2. How do DNA methylation marker profiles compare between self-sampled anal swabs and clinician-obtained anal biopsies in women with low-grade (LSIL) versus high-grade (HSIL) squamous intraepithelial lesions? Method: Women included in sub-study A who are referred to HRA/endoscopy due to hrHPV positivity will be sampled for DNA-methylation both with a self-sampled anal swab, healthcare personnel collected anal swab and with a biopsy. Quantitative Multiplex Methylation-Specific PCR method will be used to quantify the DNA methylation in host target genes including multiple target genes.

Data analysis and statistics: Correlation between self-sampled samples and biopsies will be assessed. Differences in methylation levels across the different histological categories and HPV status will be visualized using boxplots and tested for statistical significance using the Kruskal-Wallis test, followed by pairwise Mann-Whitney U-tests, with the Bonferroni correction. For evaluation of the diagnostic performance of the markers, the investigators will perform univariable mixed-effect ordinal logistic regression for the individual markers. Power calculation: A sample size of 300 women will provide the investigators with 80% statistical power (assuming α=0.05) given an expected prevalence of LSIL of at least 30% and HSIL of 25%.

ELIGIBILITY:
Inclusion Criteria:

* Women (biological sex) with HIV
* 45 years old or older
* attending the out-patient HIV departments at Karolinska University Hospital in Stockholm, the South Hospital in Stockholm, and Sahlgrenska University Hospital in Gothenburg

Exclusion Criteria:

* Women who have had anal cancer
* women who have had rectal amputation

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive anal hrHPV test | at inclusion and through study completion, an average of 1 year
  Number of participants with positive anal hrHPV test

SECONDARY OUTCOMES:
Low-grade (LSIL) and high-grade (HSIL) squamous intrepithelial lesions | at inclusion and through study completion, an average of one year
  Number of participants with Low-grade (LSIL) and high-grade (HSIL) squamous intrepithelial lesions
Circulating HPV DNA level in plasma | at inclusion and through study completion, an average of one year
  Circulating HPV DNA level in plasma
Host DNA methylation markers | at inclusion and through study completion, an average of one year
  Differences in methylation levels across the different histological categories and HPV status
Number of cases of anal cancer prevented due to screening and early treatment of HSIL | ten years
  Number of cases of anal cancer prevented due to screening and early treatment of HSIL
Number of HSIL cases detected and treated, and quality-adjusted life years gained from preventing cancer progression | four years
  Number of HSIL cases detected and treated, and quality-adjusted life years gained from preventing cancer progression
HPV ct levels | at inclusion and through study completion, an average of one year
  HPV ct levels compared to LSIL and HSIL outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Christina Carlander, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data cannot be shared due to ethical restrictions. Coding and aggregated data can be shared after publication